CLINICAL TRIAL: NCT05276297
Title: A Phase 2, Single-blinded, Randomised, Controlled Multi-country Study to Evaluate the Safety, Reactogenicity, Efficacy and Immune Response Following Sequential Treatment With an Anti-sense Oligonucleotide (ASO) Against Chronic Hepatitis B (CHB) Followed by Chronic Hepatitis B Targeted Immunotherapy (CHB-TI) in CHB Patients Receiving Nucleos(t)Ide Analogue (NA) Therapy
Brief Title: A Study on the Safety, Efficacy and Immune Response Following Sequential Treatment With an Anti-sense Oligonucleotide Against Chronic Hepatitis B (CHB) and Chronic Hepatitis B Targeted Immunotherapy (CHB-TI) in CHB Patients Receiving Nucleos(t)Ide Analogue (NA) Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 217023; 2021-003567-10 (EudraCT Number); 2024-512352-38-00 (EU CTIS Number)
Record Dates: First submitted 2022-02-14; First posted 2022-03-11 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B virus; Chronic Hepatitis B; Chronic Hepatitis B targeted immunotherapy; Bepirovirsen; Safety; Reactogenicity; Efficacy; Immunogenicity
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Who Masked: Participant
Masking Description: Open-label for Treatment 1 and single-blinded for Treatment 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ASO24-TI Group (Experimental): Eligible participants receive GSK3228836 (Treatment 1) study intervention for 24 weeks of Treatment 1 period, followed by GSK3528869A (Treatment 2) study intervention administered at Days 1, 57, 113 and 169 of Treatment 2 period. The interval between Treatment 1 and Treatment 2 is preferably 1 week, with the possibility to extend up to 12 weeks.
  Interventions: Drug: GSK3228836; Biological: GSK3528869A
- ASO24 Group (Active Comparator): Eligible participants receive GSK3228836 (Treatment 1) study intervention for 24 weeks of Treatment 1 period, followed by non-active control (Treatment 2) study intervention administered at Days 1, 57, 113 and 169 of Treatment 2 period. The interval between Treatment 1 and Treatment 2 is preferably 1 week, with the possibility to extend up to 12 weeks.
  Interventions: Drug: GSK3228836; Drug: Control
- ASO12-TI Group (Experimental): Eligible participants receive GSK3228836 (Treatment 1) study intervention for 12 weeks of Treatment 1 period, followed by GSK3528869A (Treatment 2) study intervention administered at Days 1, 57, 113 and 169 of Treatment 2 period. The interval between Treatment 1 and Treatment 2 is preferably 1 week, with the possibility to extend up to 12 weeks.
  Interventions: Drug: GSK3228836; Biological: GSK3528869A
- ASO12 Group (Active Comparator): Eligible participants receive GSK3228836 (Treatment 1) study intervention for 12 weeks of Treatment 1 period, followed by non-active control (Treatment 2) study intervention administered at Days 1, 57, 113 and 169 of Treatment 2 period. The interval between Treatment 1 and Treatment 2 is preferably 1 week, with the possibility to extend up to 12 weeks.
  Interventions: Drug: GSK3228836; Drug: Control

INTERVENTIONS:
Drug: GSK3228836 — 2 doses of GSK3228836 study intervention administered subcutaneously once per week for 12 weeks (Day 1 up to Day 78) to participants in ASO12-TI and ASO12 groups, or for 24 weeks (Day 1 up to Day 162) to participants in ASO24-TI and ASO24 groups, plus loading doses administered at Day 4 and Day 11 (2 doses each day) to participants in all groups during Treatment 1 period.
  Other Names: Bepirovirsen
Biological: GSK3528869A — The GSK3528869A chronic Hepatitis B targeted immunotherapy (CHB-TI) consisting of 4 doses administered intramuscularly as follows:
  * 1 dose of the Chimpanzee adenovectored HBV vaccine (ChAd155-hIi-HBV) at Day 1 of Treatment 2 period.
  * 1 dose of the Modified Vaccinia Virus Ankara HBV vaccine (MVA-HBV) at Day 57 of Treatment 2 period.
  * 2 subsequent doses of the AS01B-4-adjuvanted HBc-HBs proteins (HBc-HBs/AS01B-4) administered at Day 113 and Day 169 of Treatment 2 period.
  Arms: ASO12-TI Group; ASO24-TI Group
Drug: Control — 4 doses of non-active control administered intramuscularly in the deltoid region of the non-dominant arm at Days 1, 57, 113 and 169 to participants in ASO24 and ASO12 control groups during Treatment 2 period.
  Arms: ASO12 Group; ASO24 Group

SUMMARY:
This study will assess the safety, efficacy and immune response following the sequential treatment of GlaxoSmithKline's (GSK) ASO compound (GSK3228836) and CHB-TI (GSK3528869A) in participants 18 to 65 years stable on NA treatment for CHB. The aim is to quantify the efficacy of sequential therapy as well as to determine an added value of sequential therapy over GSK3228836 therapy in CHB patients treated with NAs. In addition, the study will assess the effect of different treatment durations of GSK3228836 (12 or 24 weeks) prior to initiating GSK3528869A treatment.

DETAILED DESCRIPTION:
The study follow-up period was reduced from 2 years post last dose to at least 1 year post last dose, with Visit Treatment 2-Day 505 defined as the last visit of the study. For participants who completed visits Treatment 2-Day 673 or Treatment 2-Day 841, those visits were considered the last study visit.

ELIGIBILITY:
Inclusion criteria:

* Participants, who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written or witnessed/thumb printed informed consent obtained from the participant prior to performance of any study-specific procedure.
* A male or female between, and including, 18 and 65 years of age at the time of signing of the informed consent (except for South Korea, where a male or female between, and including, 19 and 65 years of age at the time of signing of the informed consent can participate in the study).
* Participants who are Hepatitis B envelop antigen (HBeAg) positive or negative.
* Participants who have documented chronic HBV infection >=6 months prior to screening and currently stable on NA therapy defined as no changes to their nucleos(t)ide regimen from at least 6 months prior to screening and with no planned changes to the stable regimen over the duration of the study.
* CHB patient, under and adherent to treatment with a NA with high barrier to resistance (e.g. entecavir, tenofovir disoproxil fumarate and tenofovir alafenamide).
* Participants with ALT <=2x upper limit of normal (ULN) (i.e., no ALT >2x ULN) documented in approximately the last 6 months.
* Participants with plasma or serum HBsAg concentration >100 IU/mL.
* Participants must be adequately suppressed, defined as plasma or serum HBV DNA <90 IU/mL.
* A male participant is eligible if he agrees to the following during the intervention period and for at least 90 days after the last dose of study intervention:

  * Refrain from donating sperm
  * AND be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent OR Must agree to use contraception/barrier as detailed below.
  * Agree to use a male condom [and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak] when having sexual intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant.
* A female participant is eligible:

  * If she is not pregnant or breastfeeding
  * AND at least one of the following conditions applies:
  * Is not a WOCBP
  * Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency during the intervention period and for at least 90 days after the last dose of study treatment.
* A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 24 hours before the first dose of study intervention.

Exclusion criteria:

Medical conditions

* Clinically significant abnormalities, aside from chronic HBV infection.
* Co-infection with:

  * Current or past history of HCV
  * HIV
  * HDV
* History of or suspected liver cirrhosis and/or evidence of cirrhosis as determined by:

  * both AST-Platelet Index (APRI) >2 and FibroSure/FibroTest result >0.7
  * Liver biopsy (METAVIR Score F4) or Liver stiffness >12 kPa
* FibroScan TE score >9.6 kPa and FibroTest score >0.59 at Screening.
* Diagnosed or suspected HCC.
* History of:

  * malignancy within the past 5 years except of specific cancers that are cured by surgical resection
  * vasculitis or presence of symptoms and signs of potential vasculitis
  * extrahepatic disorders possibly related to HBV immune conditions
* Positive (or borderline positive) ANCA at screening.
* Low C3/C4 at screening AND evidence of past history or current manifestations of vasculitic/inflammatory/autoimmune conditions.
* History of alcohol or drug abuse/dependence.
* QTcF >=450 msec.
* Laboratory results as follows:

  * Serum albumin <3.5 g/dL
  * GFR <60 mL/min/1.73m^2
  * INR >1.25
  * PLT count <140x10^9/L
  * HGB <10 g/dl
  * T Bil >1.25xULN unless considered as clinically not significant by the Investigator
  * ACR >=0.03 mg/mg
* Medical history of hepatic decompensation.
* Planned or previous liver transplantation.
* Documented evidence of other currently active cause of hepatitis.
* Any other clinical condition that might pose additional risk to the participant due to participation in the study.
* Major congenital defects.
* Recurrent history or uncontrolled neurological disorders or seizures.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention(s).

Prior/Concomitant therapy

* Use of any investigational or non-registered product other than the study interventions within 30 days before the first dose of study interventions, or their planned use during the study.
* Use of systemic cytotoxic agents, chronic antiviral agents or Chinese herbal medicines which may have activity against HBV within 6 months prior the study.
* Currently taking, or took within 12 months of screening, any interferon-containing therapy.
* Administration of adenovirus/adenovector-based or MVA-based vaccine within the last 12 months, except for adenovirus/adenovector-based COVID-19 vaccines that could be administered up to 30 days prior to the first study vaccine dose (applicable for all patients except for the patients in France) OR Administration of adenovirus/adenovector-based or MVA-based vaccine within the last 12 months (applicable for the patients in France only).
* Planned administration/administration of a vaccine not foreseen by the study protocol within 14 days before the first dose and/or 30 days after the last dose of study intervention administration, with the exception of influenza vaccine that may be given at any time except within a 7-day period before or after each dose and COVID-19 vaccine that may be given at any time except within a 30-day period before or after each vaccine dose apart from COVID-19 mRNA based-vaccines that may be administered any time except for the period of 14 days before and 30 days after each study vaccine dose.
* Administration of:

  * long-acting immune-modifying drugs at any time during the study
  * immunoglobulins and/or any blood products or plasma derivatives within 3 months before the first dose of study interventions or planned administration during the study
* Chronic administration of immunosuppressants or other immune-modifying drugs within 3 months prior to the first study intervention (e.g. prednisone equivalent >=20 mg/day; >=10 mg/day applicable in Germany only). Inhaled and topical steroids are allowed.
* Participants for whom immunosuppressive treatment is not advised.
* Treatment with nephrotoxic drugs or competitors of renal excretion within 2 months prior to Screening or planned during the study.
* Participants requiring anti-coagulation therapies.

Prior/Concurrent clinical study experience

* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been/will be exposed to an investigational/a non-investigational intervention.
* Previous participation in clinical trials with administration of either GSK3228836 or GSK3528869A.
* Previous participation in a clinical study in which he/she has received an investigational product within the following time period prior to the first dosing day in the current study: 5 half-lives or twice the duration of the biological effect of the study treatment or 90 days.
* Prior treatment with any other oligonucleotide/siRNA within 12 months prior to the first dosing day.

Other exclusions:

* Pregnant or lactating female.
* Female planning to become pregnant/to discontinue contraceptive precautions.
* Any study personnel or their immediate dependents, family, or household members.
* History of/sensitivity to GSK3228836, or components thereof, or a history of drug or other allergy that contraindicates their participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Percentage of participants reporting any grade 3 adverse event (AE) from first dose of GSK3228836 up to study end | From first dose of GSK3228836 (Treatment 1 -Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
  An AE is any untoward medical occurrence (an unfavourable/unintended sign - including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant that is temporally associated with the study intervention. A grade 3 AE is an AE which prevents normal, everyday activities (in adults, such an AE would, for example, prevent attendance at work/school and would necessitate the administration of corrective therapy).
Percentage of participants reporting any serious adverse event (SAE) from first dose of GSK3228836 up to study end | From first dose of GSK3228836 (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or is an abnormal pregnancy outcome.
Percentage of participants reporting any adverse events of special interest (AESIs) grade 3 or higher from first dose of GSK3228836 up to study end | From first dose of GSK3228836 (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
  AESI related to GSK3228836 treatment include thrombocytopenia, alanine transaminase (ALT) increases, vascular inflammation and complement activation, renal injury or injection site reactions.
  AESI related to GSK3528869A include liver disease-related (LDR) AEs, hematological AESI or potential immune-mediated diseases (pIMDs).
  A grade 3 AE is an AE which prevents normal, everyday activities (in adults, such an AE would, for example, prevent attendance at work/school and would necessitate the administration of corrective therapy).
Percentage of participants who achieve sustained virologic response (SVR) for 24 weeks after the planned end of active treatment in the absence of rescue medication, and difference between treatment arms (corresponding to GSK3228836 regimens) | For up to 24 weeks after the planned end of active treatment (planned end of active treatment = Treatment 1-Day 78 for ASO12 group, Treatment 1-Day 162 for ASO24 group and Treatment 2-Day 169 for ASO12-TI and ASO24-TI groups)
  SVR is defined as Hepatitis B surface antigen (HBsAg) below (<) lower limit of quantification (LLOQ) and HBV deoxyribose nucleic acid (DNA) < LLOQ.
  Rescue medication is defined as any medication initiated for the purpose of antiviral suppression other than the background stable NA therapy irrespective of the reason.

SECONDARY OUTCOMES:
Percentage of participants reporting each solicited administration site event post-GSK3528869A study intervention administration | Within 7 days post-administration (day of administration + 6 subsequent days) of each dose of GSK3528869A study intervention
  The solicited administration site events include pain, redness and swelling.
Percentage of participants reporting each solicited systemic event post-GSK3528869A study intervention administration | Within 7 days post-administration (day of administration + 6 subsequent days) of each dose of GSK3528869A study intervention
  The solicited systemic events include fatigue, fever, headache, myalgia, arthralgia and chills. Fever is defined as temperature equal to or above (>=) 38.0°C/100.4°F. The preferred location for measuring temperature is the oral cavity.
Percentage of participants reporting any unsolicited AE post-GSK3528869A study intervention administration | Within 30 days post-administration (day of administration + 29 subsequent days) of each dose of GSK3528869A study intervention
  An unsolicited AE is an AE that was not included in a list of solicited events. Unsolicited events must have been spontaneously communicated by a participant who has signed the informed consent. Unsolicited AEs include both serious and non-serious AEs.
Percentage of participants reporting any AE from first dose of GSK3228836 up to study end | From first dose of GSK3228836 (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
  An AE is any untoward medical occurrence (an unfavourable/unintended sign - including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant that is temporally associated with the study intervention.
Percentage of participants reporting any AESIs from first dose of GSK3228836 up to study end | From first dose of GSK3228836 (Treatment 1-Day 1) up to the study end (Treatment 2-Day 505/Day 673/Day 841)
  AESI related to GSK3228836 treatment include thrombocytopenia, ALT increases, vascular inflammation and complement activation, renal injury or injection site reactions. AESI related to GSK3528869A include liver disease-related AEs, hematological AESIs or pIMDs.
Percentage of participants reporting any pIMDs from first dose of GSK3528869A up to study end | From first dose of GSK3528869A (Treatment 2-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
  pIMDs are a subset of AESIs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Percentage of participants reporting hematological, biochemical or urinalysis laboratory abnormalities at pre-defined time points during Treatment 1 period | At pre-defined time points during Treatment 1 period (from Treatment 1-Day 1 until Treatment 1-Day 78 for ASO12-TI and ASO12 groups, and from Treatment 1-Day 1 until Treatment 1-Day 162 for ASO24-TI and ASO24 groups)
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Percentage of participants reporting hematological, biochemical or urinalysis laboratory abnormalities at pre-defined time points during Treatment 2 period | At pre-defined time points during Treatment 2 period (from Treatment 2-Day 1 until Treatment 2-Day 199)
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Percentage of participants reporting hematological, biochemical or urinalysis laboratory abnormalities at pre-defined time points during follow-up period | At pre-defined time points during follow-up period (from Treatment 2-Day 225 until Treatment 2-Day 505/Day 673/Day 841)
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Percentage of participants who achieve quantitative Hepatitis B surface antigen assessment (qHBsAg) decrease and HBsAg loss at pre-defined time points from GSK3228836 baseline (Treatment 1-Day 1) up to study end | At pre-defined time points from GSK3228836 baseline (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
  qHBsAg decrease is defined as ≥ 0.5 log decrease and ≥ 1-log decrease. The analysis is performed by considering the HBsAg status prior to GSK3228836 as baseline.
Changes in qHBsAg at pre-defined time points from GSK3228836 baseline (Treatment 1-Day 1) up to study end | At pre-defined time points from GSK3228836 baseline (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
  Changes in serum qHBsAg from GSK3228836 baseline are expressed as geometric mean ratios (GMRs). The analysis is performed by considering the HBsAg status prior to GSK3228836 as baseline.
Percentage of participants with HBsAg loss and anti-HBs seroconversion | At pre-defined time points from first dose of GSK3228836 (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
  A participant is counted only when both HBsAg loss and anti-HBs seroconversion are reported for the participant. Seroconversion is defined as the appearance of antibodies (i.e., concentrations/titer greater than or equal to the LLOQ) in the serum of participants seronegative before GSK3528869A administration.
Geometric mean concentrations (GMCs) of qHBsAg | At pre-defined time points from first dose of GSK3228836 (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
Duration of SVR in terms of time to the first occurrence of HBsAg reversion and/or HBV DNA reversion | From Treatment 1-Day 1 up to first occurrence of HBsAg reversion and/or HBV DNA reversion, assessed from Treatment 1-Day 1 up to Treatment 2-505/Day 673/Day 841
  HBsAg reversion is defined as HBsAg >LLOQ or HBV DNA >LLOQ, confirmed by 2 consecutive visits at least 1 month apart.
Percentage of participants who experienced HBV DNA virologic breakthrough | At pre-defined time points from first dose of GSK3228836 (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
  HBV DNA virologic breakthrough is defined at 1-log increase from nadir in HBV DNA or HBV DNA becoming quantifiable after being below the LLOQ.
Percentage of participants with anti-HBc antibody response | At pre-defined time points from first dose of GSK3228836 (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
Anti-HBc antibody concentrations | At pre-defined time points from first dose of GSK3228836 (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
  Anti-HBc antibody concentrations are expressed as geometric mean concentrations (GMCs).
Percentage of participants who achieved HBsAg seroconversion | At pre-defined time points from first dose of GSK3228836 (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
  Seroconversion is defined as the appearance of antibodies (i.e., concentrations/titer greater than or equal to the LLOQ) in the serum of participants seronegative before GSK3528869A administration.
Percentage of participants with anti-HBs antibody response | At pre-defined time points from first dose of GSK3228836 (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
Anti-HBs antibody concentrations | At pre-defined time points from first dose of GSK3228836 (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
  Anti-HBs antibody concentrations are expressed as GMCs.
Percentage of participants with anti-HBs antibody concentrations equal to or above (≥) 10 mIU/mL | At pre-defined time points from first dose of GSK3228836 (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
Percentage of participants with anti-HBs antibody concentrations equal to or above (≥) 100 mIU/mL | At pre-defined time points from first dose of GSK3228836 (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
Frequency of HBc-specific CD4+ T-cells | At pre-defined time points from first dose of GSK3228836 (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
  Frequency of HBc-specific CD4+ T-cells is expressed as HBc-specific CD4+ T-cells per million peripheral blood mononuclear cells (HBc-specific CD4+ T-cells/million PBMCs).
Frequency of HBs-specific CD4+ T-cells | At pre-defined time points from first dose of GSK3228836 (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
  Frequency of HBs-specific CD4+ T-cells is expressed as HBs-specific CD4+ T-cells/million PBMCs.
Frequency of HBc-specific CD8+ T-cells | At pre-defined time points from first dose of GSK3228836 (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
  Frequency of HBc-specific CD8+ T-cells is expressed as HBc-specific CD8+ T-cells/million PBMCs.
Frequency of HBs-specific CD8+ T-cells | At pre-defined time points from first dose of GSK3228836 (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
  Frequency of HBs-specific CD8+ T-cells is expressed as HBs-specific CD8+ T-cells/million PBMCs.
Number of HBc- and HBs-specific CD4+ T cells responders | At pre-defined time points from first dose of GSK3228836 (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)
Number of HBc- and HBs-specific CD8+ T cells responders | At pre-defined time points from first dose of GSK3228836 (Treatment 1-Day 1) up to study end (Treatment 2-Day 505/Day 673/Day 841)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (41):
- GSK Investigational Site, Edegem, Belgium
- Bulgaria (4):
  - GSK Investigational Site, Sliven
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Veliko Tarnovo
  - GSK Investigational Site, Vratsa
- France (4):
  - GSK Investigational Site, Clichy
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Strasbourg
- Germany (3):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Leipzig
- GSK Investigational Site, Pokfulam, Hong Kong
- Italy (4):
  - GSK Investigational Site, Bergamo
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Rozzano MI
- Philippines (2):
  - GSK Investigational Site, Makati City
  - GSK Investigational Site, Pasig
- Poland (3):
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Mysłowice
  - GSK Investigational Site, Łańcut
- Romania (2):
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Craiova Dolj
- GSK Investigational Site, Singapore, Singapore
- Spain (5):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Vigo
- Taiwan (5):
  - GSK Investigational Site, Chiayi City
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Linkou - Taoyuan Hsien
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Tainan
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
- Turkey (Türkiye) (2):
  - GSK Investigational Site, Istanbul
  - GSK Investigational Site, Rize
- United Kingdom (2):
  - GSK Investigational Site, Cottingham
  - GSK Investigational Site, Leicester

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.